CLINICAL TRIAL: NCT00342199
Title: Epidemiological Surveillance in India of Group A Streptococcal Infections Including Pharyngitis and Impetigo Supported by Indo-US Vaccine Action Program
Brief Title: Surveillance of Streptococcal Infections in Children in India
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901190; 01-I-N190
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-02-26

CONDITIONS: Group A Beta Hemolytic Streptococcal (GAS) Infection
Keywords: Incidence; Prevalence; Immunity; Bacteriology; Pathogenesis
MeSH Terms: conditions — Infections

SUMMARY:
Information from this study is needed to plan an eventual trial of a GAS vaccine in India if and when one is available. A GAS vaccine is currently a priority of the Indian Council for Medical Research (ICMR), and this project has been approved by the Joint Working Group (US and Indian Delegates) of the Vaccine Action Program, a joint effort of the ICMR and NIAID to implement cooperative efforts between the two countries on mutual objectives in vaccine development. Currently, several GAS vaccines are in development, supported by NIAID, and other sources, and one candidate is in phase one clinical trial authorized by the FDA. Information on the antigenic structure of GAS isolated in India will be needed for planning vaccine composition. It is the view of the Indian Ministry of Health and Indian Council for Medical Research that eventual prevention and control of rheumatic fever and rheumatic heart disease in India, now a heavy burden on the children will require a GAS vaccine, which requires both access to primary health care and a vaccine if and when it is available.

Information on incidence is needed to determine the size of a future vaccine cohort in order to obtain a statistically significant result on vaccine efficacy. Although unrelated to vaccine development, information on the incidence of GAS pharyngitis is needed in India to implement primary and secondary acute rheumatic fever (ARF) and rheumatic heart disease (RHD) prevention programs as were implemented in the USA and Europe forty years ago.

A vaccine trial is not part of this study, nor is there any intervention, other than antibiotic treatment of all children volunteers who develop GAS pharyngitis or impetigo.

An additional point should be made about the importance of obtaining epidemiological data on streptococcal disease in India, and on the emm types of GAS that cause infections. The population of India is over one billion people, representing nearly twenty five percent of the world's population. Information on GAS epidemiology from India is scant to say the least, and it is sorely needed. We now know that streptococcal toxic shock syndrome and fasciitis that have occurred in the U. S., Europe, Australia, and Japan, with greater frequency in recent years are caused by several genetically similar emm types of GAS. The implication of such genetic and epidemiologic data is that these genetically related strains have spread worldwide, Current information from India is far too limited to know if these virulent strains of GAS occur in India, and if they do, to what extent might they be the cause of frequent invasive disease in hospitalized patients.

Equally important, we do not know if a potentially high virulent GAS strain is currently emerging in some locale(s) in India, and what possible threat it might become, if it were to be transported to other worldwide geographic regions. Although not a specific aim of this proposal, the surveillance conducted to accomplish the aims of this protocol will provide essential information on the possible emergence of an unexpected emm type with pathogenic potential.

...

DETAILED DESCRIPTION:
This is an epidemiological study on the incidence of Group A beta hemolytic streptococcal (GAS) infections (both pharyngitis and impetigo) in school-age children in two rural area of India: surveillance in four schools, in the north in the Punjab near Chandigarh conducted by the medical staff of the Department of Community Medicine Post-graduate Institute for Medical Research and Training (PGI); and in one school in the south in Tamil Nadu near Vellore conducted by the medical staff of the Department of Community Medicine, Christian Medical College (CMC).

Children and their teachers were questioned weekly for a history of GAS infection. On all children suspected from the history of a streptococcal infection of the pharynx or the skin, a physical examination of nose, throat, ears and skin was performed and throat culture and or skin culture and blood sample were taken for subsequent antibody determination. The diagnosis of GAS infection was made on the basis of established clinical criteria and the isolation of GAS from throat and skin lesion cultures.

The surveillance of the children was completed in March '04 in Vellore, and in April '04 in Chandigarh. For the next year, there will be extensive analysis of the clinical data; analysis of the isolated GAS for emm type and other bacteriologic characteristics; and epidemiologic analysis in a search for patterns of distribution of GAS infections by sex, age, school and session.

The general objectives have been:

To establish population-based surveillance to determine the incidence of GAS infection in school children age 7-11, to characterize the M protein of the newly isolated strains of GAS by emm gene sequencing,

1. to identify surrogate markers of protective immunity relevant to vaccine development such as serum antibody to the M type-specific peptides and cysteine protease, and
2. to define the molecular epidemiology of GAS in terms of those characteristics that are relevant to vaccine-induced immunity.

Information from this study is needed to plan an eventual trial of a vaccine(s) if and when one is available. Information on the antigenic structure of GAS isolated in India will be needed for planning vaccine composition. Information on incidence is needed to determine the size of a future cohort that will be needed to obtain a statistically significant result on vaccine efficacy.

A vaccine trial is not part of this study, nor was there any intervention, other than diagnostic procedures and antibiotic treatment of all who develop a GAS infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

All students (approximately 225-250) attending four classes in four rural schools, grades 2-5, in rural villages near Chandigarh, and all students in classes 2-6 approximately 225-250 attending one rural village school near Vellore were asked to participate.

Approximately an equal number of boys and girls participated.

Selection of the schools for the study was determined by such factors as the accessibility to a rural regional clinic, housing facilities for medical staff, and passable tertiary roads to the villages and the schools.

EXCLUSION CRITERIA:

All volunteers had a history of acute rheumatic fever and acute glomerulonephritis and evidence of rheumatic fever and rheumatic heart disease on physical examination at the initial survey were excluded from the study.

Excluded also was a child with a compromising illness such as cystic fibrosis that might require frequent or intermittent antibiotic treatment.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 663 (Actual)
Dates: Start 2001-07-03; Study Completion 2014-02-26

CONTACTS AND LOCATIONS:
Overall Officials: Dean A Follmann, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- India (2):
  - Post Graduate Institute of Medical and Experimental Research, Chandigarh
  - Christian Medical College, Vellore

REFERENCES:
- [Background] Schwartz B, Facklam RR, Breiman RF. Changing epidemiology of group A streptococcal infection in the USA. Lancet. 1990 Nov 10;336(8724):1167-71. doi: 10.1016/0140-6736(90)92777-f. PMID 1978035
- [Background] Kaplan EL. T. Duckett Jones Memorial Lecture. Global assessment of rheumatic fever and rheumatic heart disease at the close of the century. Influences and dynamics of populations and pathogens: a failure to realize prevention? Circulation. 1993 Oct;88(4 Pt 1):1964-72. doi: 10.1161/01.cir.88.4.1964. No abstract available. PMID 8403347
- [Background] Gulley RL, Fex J, Wenthold RJ. Uptake of putative neurotransmitters in the organ of Corti. Acta Otolaryngol. 1979;88(3-4):177-82. doi: 10.3109/00016487909137157. PMID 40384